CLINICAL TRIAL: NCT02687568
Title: Values of Enhanced Monitoring by EEG Recording ( Narcotrend ) as an Adjunct to Standard Monitoring for Sedation in Colonoscopy
Brief Title: Values of Enhanced Monitoring by EEG Recording (Narcotrend) for Sedation in Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Andrea Riphaus, PD Dr. Andrea Riphaus, Ruhr University of Bochum
Other Study IDs: 4439-12
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Electroencephalography; Propofol; Gender Identity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: EEG monitoring — Value of EEG monitoring as adjunct to standard monitoring

SUMMARY:
Endoscopic examinations and particularly long-lasting interventions can be uncomfortable for patients. Pain and vasovagal reactions are common. Therefore, the implementation is generally recommended under sedation and also carried out in practice here.

The vital signs monitoring to avoid complications is dictated by current national guidelines. Necessary measures of monitoring include pulse oximetry and blood pressure measurements. In patients with severe heart disease an ECG recording should be used additionally. Moreover, the guidelines require that the sedation is clinically monitored continuously to avoid an unwanted anesthetic stage. Such evaluation, however, is often difficult under clinical conditions and even counterproductive, since a constant response and tactile stimulation of the patient (to check clinically the depth level of sedation ), interrupts endoscopic complex intervention. However, clinical most relevant aspect is the avoidance of unrecognized transition of patients from the stage of deep sedation in an anesthetic stage.

Current recommendations do not take into account new study results from a gender perspective, which showed that women and men need a different wake-up time using the EEG derivation means by using the Narcotrend after total intravenous anesthesia, which may be due to different total doses of sedatives needed. However, the research group has been demonstrated in a previous study that most likely caused by the use of EEG monitoring (Narcotrend) an effective adaptation of sedation, in particular a more rapid recovery time by a lower dose of the administered sedative for a continuous sedation stage D0-D2 endoscopic retrograde cholangiopancreatography-(ERCP).

In the presented study the investigators evaluate the extent of gender differences in the wake-up time after sedation with propofol during colonoscopy when using EEG monitoring.

DETAILED DESCRIPTION:
Endoscopic examinations and particularly long-lasting interventions can be uncomfortable for patients. Pain and vasovagal reactions are common. Therefore, the implementation is generally recommended under sedation and also carried out in practice here.

In interventional and longer lasting interventions (for example colonoscopy, endoscopic ultrasonography, ERCP) as opposed to purely diagnostic examinations is often deep sedation.Use of propofol in terms of sedation efficacy and the wake-up time or quality is superior to the use of benzodiazepines (plus opiates) , while patient safety is the same.

The vital signs monitoring to avoid complications is dictated by current national guidelines. Necessary measures of monitoring include pulse oximetry and blood pressure measurements. In patients with severe heart disease an ECG recording should be used additionally. Moreover, the guidelines require that the sedation is clinically monitored continuously to avoid an unwanted anesthetic stage. Such evaluation, however, is often difficult under clinical conditions and even counterproductive, since a constant response and tactile stimulation of the patient (to check clinically the depth level of sedation ), interrupts endoscopic complex intervention. However, clinical most relevant aspect is the avoidance of unrecognized transition of patients from the stage of deep sedation in an anesthetic stage.

Current recommendations do not take into account new study results from a gender perspective, which showed that women and men need a different wake-up time using the EEG derivation means by using teh Narcotrend after total intravenous anesthesia, which may be due to different total doses of sedatives needed. However, the research group has beendemonstrated in a previous study that most likely caused by the use of EEG monitoring (Narcotrend) an effective adaptation of sedation, in particular a more rapid recovery time by a lower dose of the administered sedative for a continuous sedation stage D0-D2 endoscopic retrograde cholangiopancreatography-(ERCP).

In the presented study investigators evaluate the extent of gender differences in the wake-up time after sedation with propofol during colonoscopy when using EEG monitoring.

Included are patients who undergo diagnostic or therapeutic colonoscopy, which is performed under sedation with propofol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Clinical indication for colonoscopy

Exclusion Criteria:

* Lack of consent of the patient
* ASA (American Society of Anesthesiologists) class V
* Known Pregnancy
* Emergency investigations
* Pre-existent hypotension (RRsys <90mmHg), bradycardia (HR <50 / min), hypoxia (SaO2 <90%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included are patients which is a , diagnostic or interventional colonoscopy under sedation with propofol.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
mean recovery time after propofol sedation for colonoscopy using the EEG recording EEG monitoring at stage D0 to D2 | Immediately after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Agness Karll Laatzen, Laatzen, Germany

REFERENCES:
- [Background] Wehrmann T, Grotkamp J, Stergiou N, Riphaus A, Kluge A, Lembcke B, Schultz A. Electroencephalogram monitoring facilitates sedation with propofol for routine ERCP: a randomized, controlled trial. Gastrointest Endosc. 2002 Dec;56(6):817-24. doi: 10.1067/mge.2002.129603. PMID 12447291
- [Derived] Riphaus A, Slottje M, Bulla J, Keil C, Mentzel C, Limbach V, Schultz B, Unzicker C. Women awaken faster than men after electroencephalogram-monitored propofol sedation for colonoscopy: A prospective observational study. Eur J Anaesthesiol. 2017 Oct;34(10):681-687. doi: 10.1097/EJA.0000000000000665. PMID 28873076